CLINICAL TRIAL: NCT03070847
Title: Impact of Prophylactic Tranexamic Acid on Intra and Postoperational Bleeding Reduction in Patients Undergoing Rhinoplasty Surgery. Low (10mg/kg) and Very Low (5mg/kg) Dose Comparison
Brief Title: Low vs. Very Low Dose of Prophylactic Tranexamic Acid for Bleeding Reduction During Rhinoplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bartłomiej Wódarski (Other)
Responsible Party: Sponsor-Investigator, Bartłomiej Wódarski, MD, Centre of Postgraduate Medical Education
Organization: Centre of Postgraduate Medical Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: txa01
Record Dates: First submitted 2017-02-21; First posted 2017-03-06 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Bleeding Reduction
Keywords: tranexamic acid; rhinoplasty; bleeding reduction
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded (participant, care provider, investigator). Computer block randomisation tool will be used (randomisation.com 1 block, 50 subjects per block), 50 notes with '5 mg/kg' or '10 mg/kg' will be put into sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very low dose (Experimental): Will receive single bolus of Tranexamic acid. Dose: 5mg/kg diluted in 0,9% sodium chloride (0,9% NaCl), administered IV (in the vein), 15 min before admission to operation theatre.
  Interventions: Drug: Tranexamic Acid; Drug: Sodium Chloride
- Low dose (Active Comparator): Will receive single bolus of Tranexamic acid. Dose: 10mg/kg diluted in 0,9% sodium chloride (0,9% NaCl), administered IV (in the vein), 15 min before admission to operation theatre.
  Interventions: Drug: Tranexamic Acid; Drug: Sodium Chloride

INTERVENTIONS:
Drug: Tranexamic Acid — Dose: 5mg/kg
  Other Names: Exacyl
  Arms: Very low dose
Drug: Tranexamic Acid — Dose: 10mg/kg
  Other Names: Exacyl
  Arms: Low dose
Drug: Sodium Chloride — Tranexamic Acid would be diluted in 0,9% Sodium Chloride (0,9% NaCl) to cumulative volume of 20 ml.

SUMMARY:
The purpose of this study is to determine whether very low dose of preoperative tranexamic acid (5mg/kg) is as effective as low dose (10mg/kg) for intraoperational bleeding reduction in patients undergoing elective rhinoplasty surgery.

DETAILED DESCRIPTION:
Background

Tranexamic acid is a drug registered for bleeding prevention and reduction. It is on the World Health Organisation (WHO) 'essential drugs list'. Preoperative tranexamic acid efficacy is well proved for doses between 10 and 40 mg/kg and last years and decades publications showed that 'low dose' (10mg/kg) is as efficient as higher doses but connected with less adverse effects.

Objectives

To determine whether 5 mg/kg dose is as effective as commonly used 10mg/kg dose in intraoperational bleeding reduction.

Methodology All patients would be randomised into one of two arms - low and very low dose. Patients, investigators and caregivers would be blinded. Patients would receive intravenous bolus of tranexamic acid at 15 minutes before admission to operation theatre in a dose dependent on the study arm. General, intravenous anesthesia (total intravenous anesthesia) would be performed due to hospital standards. At the end of the surgery total blood volume and adverse effects would be noted. Surgeon would asses surgical field in the Fromm scale.

The survey is planned for a two years timespan or until 50 patients have enrolled (25 for each arm).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 y.o.
* American Society of Anesthesiologists Physical Status Classification (ASA) 1-2
* signed informed consent form after reading the information about the study and talking with one of the investigators

Exclusion Criteria:

* pregnancy
* known allergies for tranexamic acid or any other substance in Exacyl
* deep vein thrombosis
* Hormone Replacement Therapy or oral contraceptive usage
* anticoagulants usage
* obesity - BMI (body mass index) >30 kg/m2
* renal disease, as glomerular filtration rate (GFR) <60 ml/min/1,73 m*m
* seizures or epilepsy in the past

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Intraoperational bleeding | during rhinoplasty
  it would be assessed at the end of the surgery by measuring blood volume in the suction device and net weight of all surgical material. (precision balance - 2 mg)

SECONDARY OUTCOMES:
Adverse effects | during rhinoplasty and first day after surgery
  any adverse effects connected with tranexamic acid usage would be noted
surgical field assesment | during rhinoplasty
  Fromm scale of surgical field would be used
surgery length | during rhinoplasty
  surgical procedure length would be noted

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny im. prof. W. Orłowskiego w Warszawie, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No